CLINICAL TRIAL: NCT02642289
Title: Probiotics: Clinical Intervention Trial in Patients With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pablo Román López (Other)
Responsible Party: Sponsor-Investigator, Pablo Román López, PhD Student, Universidad de Almeria
Organization: Universidad de Almeria (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UAL-270415
Record Dates: First submitted 2015-12-21; First posted 2015-12-30 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Fibromyalgia
Keywords: Probiotics
MeSH Terms: conditions — Fibromyalgia | interventions — Lacteol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Probiotic1: Lactobacillus acidophilus (Experimental): Dietary Supplement: Probiotics 1. 8-week probiotic food-supplement intervention with Lactobacillus acidophilus (Daily intake: 24 millions)
  Interventions: Dietary Supplement: Lactobacillus acidophilus
- Placebo (Placebo Comparator): Inactivate substance
  Interventions: Other: Placebo
- Probiotic2: Lactobacillus Rhamnosus GG ® (Experimental): Dietary Supplement: Probiotics 2 8-week probiotic food-supplement intervention with Lactobacillus Rhamnosus (Daily intake: 24 millions)
  Interventions: Dietary Supplement: Lactobacillus Rhamnosus GG ®

INTERVENTIONS:
Dietary Supplement: Lactobacillus acidophilus — Probiotic 5000, a commercial probiotic product provided by the company "Complementos Fitonutricionales, S.L."
  Arms: Probiotic1: Lactobacillus acidophilus
Dietary Supplement: Lactobacillus Rhamnosus GG ® — Ergyphilus confort, a commercial probiotic product provided by the nutritional supplements lab "Laboratorios Nutergia"
  Arms: Probiotic2: Lactobacillus Rhamnosus GG ®
Other: Placebo — Innocuous substance
  Arms: Placebo

SUMMARY:
This study evaluates the benefits of probiotics in patients with fibromyalgia syndrome.

DETAILED DESCRIPTION:
Probiotics has demonstrated to be effective in the management of anxiety and depression. Although these results are promising, more research is needed to explore the role of probiotics to improve physical, emotional and cognitive processes in different clinical populations that are associated with altered microbiome. Thus, the main aim of the present project is to explore whether the oral intake of probiotics might provide benefits to a group of patients with fibromyalgia.

The investigators expect to found significant differences between some physical, emotional and cognitive measures assessed pre- and post-treatment demonstrating the effects of microbiota on the Central Nervous System as well as its potential as a therapeutic tool for the treatment of Fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Fibromyalgia syndrome diagnosis.
* No treatment with antibiotic.
* More than a year of diagnosis
* Agreement to participate in the study.

Exclusion Criteria:

* Severe physical disability.
* Malignancy.
* Pregnancy
* Psychiatric illnesses (eg, schizophrenia or substance abuse).
* Medication usage other than as-needed analgesics (excluding long-term narcotics).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-12; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change Scores on Working memory and attentional control | Time Frame: At baseline and 8 weeks
  Corsi task

SECONDARY OUTCOMES:
Change Scores on Body Composition | Time Frame: At baseline and 8 weeks
  Fat mass. Body fat mass. Intracellular water. Extracellular water. Fat-free mass. Total body water.
Changes Scores on Cholinergic response indicators (%) | Time Frame: At baseline and 8 weeks
Changes Scores on Heart rate variability. | Time Frame: At baseline and 8 weeks
Changes Scores on Valsalva ratio. K30/15. | Time Frame: At baseline and 8 weeks
Changes Scores on Systemic vascular resistance. | Time Frame: At baseline and 8 weeks
Change Scores on Pain | Time Frame: At baseline and 8 weeks
  Index of Widespread Pain and Symptom Severity
Change Scores on Sleep Quality | Time Frame: At baseline and 8 weeks
  Pittsburgh Sleep Quality Index Questionnaire (PSQI)
Change Scores on Quality of Life | Time Frame: At baseline and 8 weeks
  The assessment of Quality of Life (SF-36)
Change Scores on Depression | Time Frame: At baseline and 8 weeks
  The Beck inventory for depression
Change Scores on Stress | Time Frame: At baseline and 8 weeks
  Determination of cortisol in urine
Change Scores on Anxiety | Time Frame: At baseline and 8 weeks
  The State-Trait Anxiety Inventory (STAI)
Change Scores on Impulsivity | Time Frame: At baseline and 8 weeks
  The Two-choice task

CONTACTS AND LOCATIONS:
Overall Officials: Angeles Fernandez, PhD, Principal Investigator — Universidad de Almeria
Locations (1):
- Pablo Roman, Almería, Almeria, Spain